CLINICAL TRIAL: NCT02345213
Title: A Post-Marketing Clinical Study of Aricept in Patients With Dementia With Lewy Bodies (DLB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2020-J081-419
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2017-12

CONDITIONS: Dementia, Lewy Body; Lewy Body Disease
Keywords: DLB; Dementia with Lewy bodies; Lewy Body Disease; Dementia; E2020; Donepezil; Aricept
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E2020 (Experimental): Treatment period: Weeks 1-2 E2020 3 mg, Weeks 3-6 E2020 5 mg, Weeks 7-12 E2020 10 mg.
  Extension period: Weeks 1-6 E2020 10 mg, After Week 7 up to week 60 E2020 10 mg.
  Interventions: Drug: E2020
- Placebo (Placebo Comparator): Treatment period: Weeks 1-12 placebo
  Extension period: Weeks 1-2 E2020 3 mg, Weeks 3-6 E2020 5 mg, After Week 7 up to week 60 E2020 10 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2020 — E2020 tablets will be orally administered once daily after breakfast
  Arms: E2020
Drug: Placebo — Matching placebo tablets will be orally administered once daily after breakfast
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy of Aricept in patients with dementia with Lewy bodies (DLB).

ELIGIBILITY:
Inclusion Criteria

1. Patients diagnosed with probable DLB according to the diagnostic criteria for DLB
2. Patients having caregivers throughout the study who submit written consent to cooperate with this study, can routinely stay with patients at least 3 days a week (at least 4 hours a day), provide patients' information necessary for this study, assist treatment compliance, and escort the patients on required visits to study institution
3. Clinical Dementia Rating (CDR) score is greater than or equal to 0.5
4. Mini-Mental State Examination (MMSE) score is greater than or equal to 10 and less than or equal to 26

Exclusion Criteria

1. Patients diagnosed with Parkinson's disease with dementia (PDD)
2. Patients who have received anti-dementia drug therapy within 12 weeks before the start of the observation period
3. Patients with a complication of serious neuropsychiatric disease(s) such as stroke, brain tumor, schizophrenia, epilepsy, normal pressure hydrocephalus, mental retardation, brain trauma with unconsciousness, or a history of brain surgery causing unrecovered deficiency
4. Patients with severe extrapyramidal disorders (Hoehn and Yahr staging score is greater than or equal to IV)
5. Patients whose systolic blood pressure is less than 90 mmHg or pulse rate is less than 50 beats/minute at screening test

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Clinician's Interview-Based Impression of Change, Plus Caregiver Input Version (CIBIC-plus) | Up to 12 weeks
  CIBIC plus is a clinician's interview-based impression of change plus the caregiver's input. It is a seven-point categorical assessment scale for evaluating global clinical function, ranging from "markedly improved" to "markedly worse".

CONTACTS AND LOCATIONS:
Overall Officials: Megumi Ohdake, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (1):
- Saitama, Japan